CLINICAL TRIAL: NCT03870451
Title: Cryocompression for Bortezomib-Induced Peripheral Neuropathy Among Multiple Myeloma Patients
Brief Title: Cryocompression Therapy for Peripheral Neuropathy in Patients With Multiple Myeloma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00056641; NCI-2019-01261 (Other: National Cancer Institute); WFBCCC 01119 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2019-03-05; First posted 2019-03-12 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cohort 1 VascuTherm5 vascular compression device (Experimental): VascuTherm5 vascular compression device Cohort 1 - Grade 2-3 neuropathy - Patients with established neuropathy (e.g. previously received bortezomib-based chemotherapy and have clinically documented CTCAE grade 2 or 3 neuropathies. Patients undergo home cryocompression therapy treatments using VascuTherm device on their non-dominant hand and foot over 30 minutes daily for 8 weeks.
  Interventions: Device: VascuTherm5 vascular compression device
- Cohort 2 VascuTherm5 vascular compression device (Experimental): VascuTherm5 vascular compression device Cohort 2 Grade 1-2 Neuropathy - Patients with new-onset neuropathy (e.g. currently receiving bortezomib-based chemotherapy have clinically documented CTCAE grade 1 or grade 2 neuropathy to explore its role in preventing worsening of CIPN in patients receiving neurotoxic chemotherapy. Patients undergo home cryocompression therapy treatments using VascuTherm device on their non-dominant hand and foot over 30 minutes daily for 8 weeks.
  Interventions: Device: VascuTherm5 vascular compression device

INTERVENTIONS:
Device: VascuTherm5 vascular compression device — VascuTherm5 vascular compression unit to function as an intermittent external pneumatic compression device

SUMMARY:
This trial studies how well cryocompression therapy works in reducing bortezomib-induced peripheral neuropathy in patients with multiple myeloma. Peripheral neuropathy (nerve pain or tingling in hands or feet) is a common side effect of chemotherapy such as bortezomib that affects the quality of life and amount of chemotherapy that can be given to many cancer patients. Cryocompression is a treatment where a glove and a boot are worn to cool down the skin. This cooling treatment is safe and does not interfere with chemotherapy treatment. Daily cryocompression therapy may reduce neuropathy caused by bortezomib chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of daily cryocompression therapy in multiple myeloma patients with bortezomib-induced peripheral neuropathy (BIPN).

SECONDARY OBJECTIVES:

I. To examine the change in patient-reported assessment of neuropathy based on the sensory, motor and autonomic neuropathy scores on the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Cancer-Induced Peripheral Neuropathy (CIPN20) (patient-reported outcome [PRO]) from baseline to 4 and 8 weeks after the start of cryocompression therapy.

II. To examine the change in physician graded assessment of peripheral neuropathy by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 criteria from baseline to 4 and 8 weeks after the start of cryocompression therapy.

III. To assess the effect on sensory and motor nerve function via nerve conduction study (NCS) (e.g. conduction velocity, latency, and amplitude) and neuro-ultrasound after 8 weeks of daily cryocompression therapy.

EXPLORATORY OBJECTIVES:

I. To explore the effect of 8 weeks of cryocompression on changes in digital artery perfusion as measured by ultrasound (US).

II. To examine the associations among the peripheral nerve assessment measures (nerve conduction and peripheral nerve US) with the patient reported outcomes (EORTC QLQ-CIPN20, PRO-CTCAE) at baseline, week 4, week 8, and for the change from baseline to week 8.

OUTLINE:

Patients undergo home cryocompression therapy treatments on their non-dominant hand and foot over 30 minutes daily for 8 weeks.

After completion of cryocompression therapy, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed multiple myeloma (any International Staging System [ISS] stage).
* Clinical symptoms of bortezomib-induced peripheral neuropathy as measured by the NCI-CTCAE.

Cohort 1: Patients with clinically documented CTCAE grade greater than or equal 2 neuropathy.

Cohort 2: Patients with clinically documented CTCAE grade 1-2 neuropathy.

• Currently or previously received bortezomib-containing regimen

Cohort 1: Patients who have previously received a bortezomib-containing regimen and have clinically documented neuropathy that is attributed to the bortezomib containing regimen.

Cohort 2: Patients who are currently receiving a bortezomib-containing regimen and have clinically documented neuropathy that is attributed to the bortezomib containing regimen.

* Age must be greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) =< 4.
* Life expectancy >= 6 months.
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document.

Exclusion Criteria:

* Self-reported or documented history of pre-existing peripheral neuropathy prior to initiation of bortezomib therapy.
* Other explanatory etiology for neuropathy.
* Presumptive evidence of congestive heart failure.
* Current deep vein thrombosis or pulmonary embolism (diagnosed within the past 6 months).
* Current pulmonary edema.
* Unable to provide accurate medical history.
* Pregnant women are excluded from this study because they will not be receiving myeloma standard of care (SOC) therapy or bortezomib-based therapy per inclusion criteria.
* Current or previously documented inflammatory phlebitis; thrombophlebitis; decompensated cardiac insufficiency; arterial dysregulation; erysipelas; carcinoma or carcinoma metastasis in the affected extremity; decompensated hypotonia; venous or arterial occlusive disease; or Raynaud's disease;
* Current monoclonal gammopathy of undetermined significance (MGUS), Waldenstroms macroglobulinemia, or Castleman disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Feasibility - Ability to complete daily 30-minute cryocompression treatments | Baseline up to 8 weeks of cryocompression therapy
  The primary outcome measure will be feasibility of daily 30-minute cryocompression treatments with a target of 60% compliance. Compliance will be measured by VCU recorded data. Patient study treatment diary will be compared and when discrepancies exist, resolved either by asking the patient or discussing with the study principal investigator. Compliance is defined as completion of 60% of prescribed treatment days. Completion of at least 25 of 30 minutes on each day will be considered completion of therapy on the prescribed day.
  Analyses will be primarily descriptive to estimate variances and effect sizes for future work. The proportion of compliance and its 95% confidence interval will be calculated for each cohort.

SECONDARY OUTCOMES:
EORTC QLQ-CIPN20 Questionnaire | Baseline up to 8 weeks of cryocompression therapy
  Chemotherapy-induced peripheral neuropathy (CIPN) is characterized by numbness, tingling, and shooting/burning pain. Patient-reported assessment of neuropathy based on sensory, motor and autonomic neuropathic pain scores (scale of 1 to 4) 1 being "not at all" and 4 being "very much." EORTC QLQ-CIPN20 (PRO) will be done at baseline, and at 4 and 8 weeks of cryocompression therapy.
NCI-CTCAE v5.0 Severity Grade Changes | Baseline up to 8 weeks of cryocompression therapy
  Physician graded assessment of peripheral neuropathy as measured by NCI-CTCAE v5.0 criteria. The CTCAE displays Grades 1 through 5 (1 = mild, 5 = death)
Change in Motor Nerve Function | Baseline and after 8 weeks of cryocompression therapy
  Tibial motor response will include tibial amplitude (mV), latency (sec) and conduction velocity (m/sec). Sural sensory response will include amplitude (mV) and latency (sec). Scores include N(normal), INC(increased), DEC(decreased), A(absent), or NA (not available)
Change in Sensory Response | Baseline and after 8 weeks of cryocompression therapy
  Sural sensory response will include amplitude (mV) and latency (sec). Scores include N(normal), INC(increased), DEC(decreased), A(absent), or NA (not available)

OTHER OUTCOMES:
Velocity changes of digital artery perfusion | Baseline and after 8 weeks of cryocompression therapy
  Pre-treatment and post-treatment velocity measurements (cm/s) will be measured by ultrasound at baseline and after 8 weeks of cryocompression therapy.
Proportion of Changes in Peripheral Nerve Function | Baseline up to 8 weeks of cryocompression therapy
  The peripheral nerve assessment measures with the patient reported outcomes (EORTC QLQ-CIPN20, PRO-CTCAE) at baseline, week 4, week 8, and for the change from baseline to week 8. Pain scores (scale of 1 to 4) 1 being "not at all" and 4 being "very much."

CONTACTS AND LOCATIONS:
Overall Officials: Roy Strowd, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT03870451/ICF_000.pdf